CLINICAL TRIAL: NCT03656679
Title: A Comparison of the Paravertebral Block Versus Pectoralis Block in Controlling Bilateral Post-mastectomy Pain in Setting of Tissue Expander Placement
Brief Title: Paravertebral Versus Pectoralis Block for Post Mastectomy Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient participant population per COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0579; NCI-2018-01743 (Other: NCI); UW17141 (Other: UWCCC); A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY/ANESTHESIO (Other: UW Madison); Protocol Version 9/12/2019 (Other: UW Madison)
Record Dates: First submitted 2018-08-17; First posted 2018-09-04 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Pain, Postoperative; Post-Mastectomy Chronic Pain Syndrome; Opioid Use
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Assessor will be provided with de-identified data for analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pectoralis Blockade(PECs) (Active Comparator): Participants undergo pectoralis nerve block (PEC II) will received anesthesia between the pectoralis major and minor in the chest while lying flat.
  Interventions: Procedure: Pectoralis Blockade (PECs)
- Paravertebral Blockade (PVB) (Active Comparator): Participants undergoing paravertebral nerve block (PVB) consisting of receiving anesthesia in the back while sitting upright.
  Interventions: Procedure: Paravertebral Blockade

INTERVENTIONS:
Procedure: Pectoralis Blockade (PECs) — Ten milliliters of 0.25% bupivacaine with 2.5 mcg/ml epinephrine will be deposited between the pectoralis major and minor (PECs I) and 20 cc of 0.25% bupivacaine with 2.5mcg/ml epinephrine deposited between the pectoralis minor and serratus anterior muscle.
  Arms: Pectoralis Blockade(PECs)
Procedure: Paravertebral Blockade — 10cc of 0.25% bupivacaine with 2.5 mcg/ml epinephrine will be deposited at two levels (T3 and T5) per side while in the sitting position.
  Arms: Paravertebral Blockade (PVB)

SUMMARY:
Post-mastectomy pain affects more than half of patients undergoing the procedure and can last for years. It has been well established that development of chronic pain is related to experienced pain in the perioperative period. This study therefore aims to assess if both acute and chronic post-operative mastectomy pain can be better managed by a novel regional anesthesia nerve block known as the pectoralis block (PECs). The PECs block is easier for patients to position for placement, has less risk of harm to nearby structures, and less risk for systemic uptake of local anesthetic in comparison to the paravertebral block. The PECs block has a strong safety profile. Standard of care at University of Wisconsin (UW) hospital is to utilize regional anesthesia for post op pain management. While PVB is performed on a regular basis at UW per surgeon request, Surgeon can request for PECS block in patients where a PVB was contraindicated (ie. coagulation issues). PECS is in fact the standard of care at other hospitals. This study will assess outcomes in the post anesthetic care unit (PACU), post-operative day 1, 7 and 30.

DETAILED DESCRIPTION:
Post-mastectomy pain occurs in up to 55% of patients and can last for months. The development of chronic pain is related to experienced perioperative pain. The development of chronic pain is related to experienced perioperative pain. There is great potential to enhance the quality of life for breast surgery patients if the hospital can improve our perioperative pain prevention techniques. New to the spectrum of multimodal analgesia is the pectoralis block (PECs), which provides anesthesia to the anterior and anterior lateral chest wall as well to the axilla. This study is about aims to compare the pectoralis block to paravertebral block with benefits of ease placement, less risk for harm to nearby structures including pneumothorax, spinal cord trauma, sympathetic block and hypotension.

Literature reveals that the pectoralis block has provided improved pain scores as well as decreases post-operative nausea and vomiting, longer block duration, and subsequent pain relief in patient. Despite these promising preliminary studies, there remains a paucity on the effectiveness of the PECs Block, particularly regarding long term outcomes for patients.

Furthermore, there is no literature to date which has evaluated the best regional anesthetic technique for patients who receive breast tissue expanders, which can cause a significant amount of muscle pain and spasm due to the intended muscle disruption during surgical placement. The primary outcomes of this study is to compare total opioid consumption during the post-surgical period limited to 24 hrs beginning at PACU admission between patients who receive bilateral pectoralis plane versus bilateral paravertebral blocks and subsequently undergo bilateral mastectomy with tissue expanders.

The secondary outcomes includes post-operative pain scores on PACU arrival and discharge, post-operative days (POD) 1, 7, and 30, presence/absence of axillary pain, muscle relaxant consumption, presence of severity of muscle spasm, total antiemetic consumption 24-hrs beginning at PACU admission, presence of chronic opioid use (Defined as consumption at 30 days), time to perform block, and PACU duration.

ELIGIBILITY:
Inclusion Criteria:

* The clinical decision has been made that the patient will have a bilateral mastectomy with tissue expander placement
* The participant is ≥ 18 years and ≤ 80 years
* Weight ≥ 60 kg and ≤ 90 kg
* The participant's primary anesthesia care team has planned for general anesthesia
* The participant agrees to receive a regional block
* American Society of Anesthesiologists class 1-3

Exclusion Criteria:

* 18 years of age or >80 years of age
* < 60 kg or > 90 kg
* Non-English speaking
* Known or believed to be pregnant
* Participant is a prisoner
* Participant has impaired decision-making capacity per discretion of the Investigator
* Standard contraindications to regional blocks (coagulopathy including abnormal INR after discontinuation of warfarin, baseline INR (international normalized ratio) >1.5, platelets <100,000, elevated PTT (prothrombin time), failure to discontinue anticoagulant medication, or infection at site)
* Significant renal, cardiac or hepatic disease per discretion of the investigator
* A clinical decision made that indicates need for a partial or complete axillary node dissection
* American Society of Anesthesiologists class 4-5
* Known hypersensitivity and/or allergies to local anesthetics
* Chronic Opioid Use (daily or almost daily use of opioids for > 3 months)
* Participant refusal

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Total Opioid Consumption | 24 hours
  Primary outcome will be total opioid consumption in 24 hours for Paravertebral Nerve Block vs. Pectoralis Nerve Block.

SECONDARY OUTCOMES:
time to perform the block | 4 hours
  To compare the following perioperative variables (pre/intraoperative): time to perform the block.
Pain score | 30 days
  To compare the following perioperative variables: pain score at time of PACU, POD 1, 7 and 30
Location of most severe pain | 30 days
  To compare the following perioperative variables location of most severe pain at PACU, POD 1, 7 and 30
Presence or absence of axillary pain | 30 days
  To compare the following perioperative variables: presence or absence of axillary pain at PACU, POD 1, 7 and 30
Presence and severity of muscle spasm | 30 days
  To compare the following perioperative variables :
  presence and severity of muscle spasm at PACU, POD 1, 7 and 30
Total muscle relaxant consumption | 30 days
  To compare the following perioperative variables: total muscle relaxant consumption at PACU, POD 1, 7 and 30
Total antiemetic consumption | 48 hours
  To compare the following perioperative variables: total antiemetic consumption at PACU and POD 1
Time in PACU and hospital duration | 48 hours
  To compare the following perioperative variables :
  time in PACU and hospital duration
Opioid consumption at POD 7 and 30 | 30 days
  To compare the following perioperative variables : Opioid consumption at POD 7 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Wilson, MD, Principal Investigator — Anesthesiology Department, University of Wisonsin Hospital and Clinics, Madison, Wisconsin, United States,53792.
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No